CLINICAL TRIAL: NCT03892174
Title: Cytokine REmoval in CRitically Ill PAtients Requiring Surgical Therapy for Infective Endocarditis (RECReATE) - an Investigator-initiated Prospective Randomized Controlled Clinical Trial Comparing Two Established Clinical Protocols
Brief Title: Cytokine REmoval in CRitically Ill PAtients Requiring Surgical Therapy for Infective Endocarditis (RECReATE)
Acronym: RECREATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Jörg Schefold, Principal Investigator, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECREATE
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Endocarditis; Sepsis; Septic Shock
MeSH Terms: conditions — Endocarditis; Sepsis; Shock, Septic | interventions — Clinical Protocols; Adsorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment protocol without adsorption (No Intervention)
- Treatment protocol with adsorption (Active Comparator)
  Interventions: Other: Treatment protocol with adsorption

INTERVENTIONS:
Other: Treatment protocol with adsorption — Adsorption while patients are in the OR on the extracorporeal circuit
  Arms: Treatment protocol with adsorption

SUMMARY:
Infectious endocarditis (IE) and other severe infections are well-known to induce significant changes in the immune response including immune functionality in a considerable number of affected patients. In fact, numerous patients with IE develop a persistent functional immunological phenotype that can best be characterized by a profound anti-inflammation and/or functional anergy. This was previously referred to as "injury-associated immunosuppression (IAI)" by Pfortmüller et al., published in Intensive Care Medicine Experimental 2017. IAI can be assessed by measurement of cellular (functional) markers. Persistence of IAI is associated with prolonged ICU length of stay, increased secondary infection rates, and death. Immunomodulation to reverse IAI was shown beneficial in immunostimulatory (randomized controlled) clinical trials. CytoSorb® treatment is currently used as standard of care in some institutions in surgically treated IE patients. The investigators aim to investigate two accepted treatment protocols and aim to explore whether adsorption with a cytokine adsorption filter can increase immune competence in treated individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for routine cardiac surgery for infectious endocarditis (diagnosed according to the predefined "DUKE" criteria) with antibiotic therapy for ≤ 14 days.
* Presence of informed consent
* Age ≥18 yrs.

Exclusion Criteria:

* Previous treatment (last 6 months) with immunologically-active biologicals or specific immunomodulatory drugs (e.g. Rituximab)
* high-dose chronic (i.e. before onset of infectious endocarditis) steroid medication with prednisone equivalent of >30 mg/d
* Patients on Extracorporeal membrane oxygenation (ECMO), or any other (pre-operative) cardiac assist device
* Moribund patient (life expectancy <14 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quantitative expression of monocytic Human Leukocyte Antigen (mHLA)-DR expression (Antibodies per cell on Cluster of Differentiation (CD)14+ monocytes/macrophages, assessed using a quantitative standardized assay) | From baseline (pre-OR, t1) to day 1 post-OR (t3)

SECONDARY OUTCOMES:
Change in mHLA-DR from baseline (pre-OR) to post-Or and 3 days post-Or. | Baseline (pre-OP) to post-OR and 3 days post-Or
  Course of mHLA-DR
Area under the curve of quantitative mHLA-DR expression | Between baseline (pre-OR), post-OR, and day 1 and 3 post-OR (multiple assessments).
  Area under the curves mHLA-DR
Change in inflammatory markers including cytokines (Interleukin (IL)-6, IL-10, C-reactive protein, White blood cell count, multiplex Enzyme linked immunosorbent assay, and inflammatory prohormones) | From baseline (pre-OR) to post-OR, and day 1 and 3 post-OR
  Change in inflammatory parameters
Change in organ dysfunction (Sepsis-related organ failure (SOFA) scores incl. subscores and Simplified acute physiology score (SAPS II scores) daily | 7-day timeframe (starting from ICu admission, assessed at day 90)
  Course of organ dysfunction
Length of ICU and hospital stay (days after surgical intervention). | Number of days on ICU and in hospital (assessed at day 90)
  Length of stay
Cumulative Therapeutic Intervention Scoring System (TISS) points (resource need) until ICU-discharge | Total number of TISS points on ICU (cumulative), assessed at day 90
  Resource use
Total amount of infused volume/transfusions on ICU | 90 days
  Need for fluid therapy
Duration of vasoactive drug therapy | 90 days
  Vasopressor use
Duration of invasive mechanical ventilation | 90 days
  Use of organ support therapy (number of days on mechanical ventilation)
ICU mortality rate | ICU stay (assessed at day 90)
  Number of non-surviving patients in both study groups
Hospital mortality rate | hospital stay (assessed at day 90)
  Number of non-surviving patients in both study groups
28 day mortality rate | 28 days beginning from ICU admission (assessed at day 90)
  Number of non-surviving patients in both study groups
90 day mortality rate | 90 days beginning from ICU admission (assessed at day 90)
  Number of non-surviving patients in both study groups
Duration of renal replacement therapy | 90 days
  Use of organ support therapy (number of days on renal replacement therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Englberger, MD, Study Director — Inselspital, Bern University Hospital
Locations (1):
- Dept of Intensive Care Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gisler F, Spinetti T, Erdoes G, Luedi MM, Pfortmueller CA, Messmer AS, Jenni H, Englberger L, Schefold JC. Cytokine Removal in Critically Ill Patients Requiring Surgical Therapy for Infective Endocarditis (RECReATE): An Investigator-initiated Prospective Randomized Controlled Clinical Trial Comparing Two Established Clinical Protocols. Medicine (Baltimore). 2020 Apr;99(15):e19580. doi: 10.1097/MD.0000000000019580. PMID 32282706